CLINICAL TRIAL: NCT01002183
Title: Evaluation of Fosmidomycin and Clindamycin When Administered Concurrently to Adult Subjects With Acute Uncomplicated Plasmodium Falciparum Malaria
Brief Title: Fosmidomycin With Clindamycin or With Clindamycin Plus Artesunate
Acronym: JP015
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Drug combination is no longer pursued
Sponsor: Jomaa Pharma GmbH (Industry)
Collaborators: Mahidol University (Other); Thammasat University (Other)
Responsible Party: Dr David BA Hutchinson, Jomaa Pharma GmbH
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JP015
Record Dates: First submitted 2009-10-26; First posted 2009-10-27 (Estimated); Last update posted 2011-09-27 (Estimated); Status verified 2010-08

CONDITIONS: Malaria
Keywords: Malaria; Plasmodium falciparum; acute uncomplicated
MeSH Terms: conditions — Malaria; Malaria, Falciparum | interventions — fosmidomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- single arm (No Intervention): Fos-clin/Arte
  Interventions: Drug: Fosmidomycin

INTERVENTIONS:
Drug: Fosmidomycin — 450 mg capsules, every 12 hrs for 3 days

SUMMARY:
The aim of this study is to evaluate the role of clindamycin and artesunate as possible combination partners for fosmidomycin to protect it from its susceptibility to recrudescent infections when used as monotherapy for acute Plasmodium falciparum malaria while retaining its excellent safety profile

DETAILED DESCRIPTION:
The scientific rationale for the use of this combination is to inhibit the ability of the parasite to synthesise isoprenoids, as precursors of many essential compounds including sterols, carotenoids and ubiquinones. This is effected through blockade of the non-mevalonate pathway by fosmidomycin as a potent inhibitor of 1-deoxy-D-xylulose 5-phosphate reductoisomerase coupled with targeting of protein biosynthesis by azithromycin through binding to the 50S ribosomal subunit. This mode of action contrasts with the ability of the human host to utilise the mevalonate pathway for isoprenoid synthesis and accounts for the safety profiles of both drugs through the mechanism of selective toxicity. Moreover it affords protection against cross resistance with existing chemotherapeutic agents.

ELIGIBILITY:
Inclusion Criteria:

* male and female subjects aged 15 to 55 years
* body mass index ≥ 18.5kg/M2
* uncomplicated P falciparum malaria with acute manifestations
* asexual parasitaemia between 500uL and 100,000uL
* ability to tolerate oral therapy
* able to give informed signed consent

Exclusion Criteria:

* signs of severe malaria, according to WHO criteria
* body mass index ≤ 18.5kg/M2
* pregnancy by history or by positive urine test
* lactation
* mixed plasmodial infection
* concomitant disease masking assessment of response, including diabetes,
* uncontrolled hypertension, heart failure, hepatic dysfunction (alanine-amino transferase >150 U/L), renal impairment (creatinine >125umol/L or 3mg/dl)
* haemoglobin < 8g/dl
* white cell count > 12000/uL
* anti-malarial treatment within previous 28 days
* symptomatic AIDS

Ages: 15 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)

PRIMARY OUTCOMES:
Efficacy of fosmidomycin and clindamycin/artesunate when co-administered to adults with acute uncomplicated P.f. malaria. | 12 months

SECONDARY OUTCOMES:
To determine the viability and infectivity of gametocytes induced by the co-administration of fosmidomycin with clindamycin or with clindamycin plus artesunate to adult subjects with acute uncomplicated Plasmodium falciparum malaria. | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Mahidol University, Bangkok, Thailand